CLINICAL TRIAL: NCT03092024
Title: Feasibility Trial of an Internet-based Exercise Program to Improve Hand Function in Patients With Scleroderma: A Scleroderma Patient-centered Intervention Network (SPIN) Study
Brief Title: Scleroderma Patient-centered Intervention Network (SPIN) Hand Program Feasibility Study
Acronym: SPIN-HAND-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Professor, Faculty of Medicine, McGill University Senior Investigator, Lady Davis Institute for Medical Research, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CODIM-MBM-12-123B
Record Dates: First submitted 2017-03-02; First posted 2017-03-27 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Systemic Sclerosis; Scleroderma; Hand; Intervention; Exercise
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIN-HAND program (Experimental)
  Interventions: Other: SPIN-HAND program
- Not Offered the SPIN-HAND program (No Intervention): Treatment as usual

INTERVENTIONS:
Other: SPIN-HAND program — The internet-based SPIN-HAND program consists of 4 modules (1) Thumb Flexibility and Strength (3 exercises); (2) Finger Bending (3 exercises); (3) Finger Extension (3 exercises); and (4) Wrist Flexibility and Strength (2 exercises). The program includes sections on developing a personalized program, goal-setting strategies and examples, progress tracking, sharing goals and progress with friends and family, and patient stories of experiences with hand disability and hand exercises. Instructional videos demonstrate and explain how to perform each exercise properly with pictures to illustrate common mistakes. Separate versions of each exercise are available for patients with mild/moderate and more severe hand involvement.
  Arms: SPIN-HAND program

SUMMARY:
The Scleroderma Patient-centered Intervention Network (SPIN) is an organization established by researchers, health care providers, and people living with scleroderma from Canada, the USA, and Europe. The objectives of SPIN are (1) to assemble a large cohort of scleroderma patients to complete outcome assessments regularly in order to learn more about important problems faced by people living with scleroderma and (2) to develop and test a series of internet-based interventions to help patients manage aspects of scleroderma, including hand limitations.

In the SPIN-HAND feasibility trial, SPIN Cohort participants with at least mild hand function limitations and an indicated interest in using an online hand exercise program will be randomized to be offered the SPIN hand exercise program or to usual care only. The core SPIN hand exercise program consists of 4 modules that address specific aspects of hand function, including Thumb Flexibility and Strength; Finger Bending; Finger Extension; and Wrist Flexibility and Strength. The program also integrates tools to support key components of successful self-management programs, including goal-setting.

The aim of the SPIN-HAND feasibility study is to collect data to assess the feasibility of the steps that need to take place as part of the main trial; required resources; and scientific aspects (e.g., withdrawal rate, outcomes measures). Data will be used to determine whether it is feasible to carry out the main study or whether changes need to be made before conducting a full-scale RCT of the SPIN-HAND program.

DETAILED DESCRIPTION:
The SPIN Cohort currently currently includes over 1700 patients from 36 sites in Canada, the USA, France, and the United Kingdom. It is anticipated that the Cohort will grow to approximately 2,000 patient by the end of 2017. SPIN Cohort patients complete outcome measures via the internet upon enrolment and subsequently every 3 months. SPIN utilizes the cohort multiple RCT (cmRCT) design as a framework for conducting trials of interventions. SPIN Cohort patients consent to allow personal data to be used for observational research, to assess intervention trial eligibility and, if eligible, be randomized. Patients also consent that if eligible and randomized to usual care, the patient's data can be used to evaluate intervention effectiveness without the patient being notified that the patient has been randomized to the usual care group and not offered the intervention. Thus, in SPIN trials, trial status is masked for patients in the control arm, who are not aware that they are in the trial, but not patients in the intervention arm. The investigative team does not interact with patients for care provision or outcome assessment, which are done automatically via the internet.

The SPIN-HAND feasibility study is embedded in the SPIN Cohort and will evaluate the feasibility of conducting full-scale RCT on the SPIN-HAND exercise program. Investigators will randomize 36-40 SPIN Cohort patients with at least mild hand function limitations and an indicated interest in using an online hand exercise program to be offered the hand exercise program or usual care only.

Randomization will occur at the time of patients' regular SPIN Cohort assessments. Eligible patients, based on questionnaire responses, will be randomized automatically using simple 1:1 randomization, using a feature in the SPIN Cohort platform, which provides immediate randomization and complete allocation sequence concealment.

Feasibility outcomes include patient eligibility and recruitment and numbers and percentages of patients who do not respond to follow-up measures. Use of the internet intervention will be described by presenting the frequency of logins and time spent on the SPIN-HAND program. Analysis of outcome measures will include the completeness of data and presence of floor or ceiling effects. Descriptive statistics will be used to provide means and standard deviations for the measures. Qualitative information and information related to management and usability of the SPIN-HAND program will inform any necessary changes to the intervention or trial procedures.

ELIGIBILITY:
Inclusion Criteria:

* SPIN Cohort patients must have a systemic sclerosis (SSc) diagnosis based on 2013 American College of Rheumatology/European League Against Rheumatism criteria confirmed by a SPIN physician, be ≥18 years old, be able to give informed consent, and be fluent in English or French.
* For the feasibility trial, eligible patients will be able to use the online intervention in English, have at least mild hand function limitations (Cochin Hand Function Scale ≥ 3) and have indicated high interest in using an online hand exercise intervention (≥7 on 0-10 scale).

Exclusion Criteria:

* Patients not able to access or respond to questionnaires via the internet are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD, PhD, Principal Investigator — Hôpital Cochin, Paris, France; Serge Poiraudeau, MD, PhD, Principal Investigator — Hôpital Cochin, Paris, France; Brett Thombs, PhD, Principal Investigator — Lady Davis Institute, Montreal, Quebec, Canada
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request

REFERENCES:
- [Derived] Kwakkenbos L, Carrier ME, Welling J, Turner KA, Cumin J, Pepin M, van den Ende C, Schouffoer AA, Hudson M, van Breda W, Sauve M, Mayes MD, Malcarne VL, Nielson WR, Nguyen C, Boutron I, Rannou F, Thombs BD, Mouthon L; SPIN Investigators. Randomized feasibility trial of the Scleroderma Patient-centered Intervention Network hand exercise program (SPIN-HAND). PeerJ. 2022 Aug 4;10:e13471. doi: 10.7717/peerj.13471. eCollection 2022. PMID 35945943
- [Derived] Carrier ME, Kwakkenbos L, Boutron I, Welling J, Sauve M, van den Ende C, Schouffoer AA, Hudson M, Thombs BD, Mouthon L; SPIN Investigators*. Randomized feasibility trial of the Scleroderma Patient-centered Intervention Network hand exercise program (SPIN-HAND): Study protocol. J Scleroderma Relat Disord. 2018 Feb;3(1):91-97. doi: 10.5301/jsrd.5000263. Epub 2017 Oct 16. PMID 35382119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessment of trial eligibility occurred during participants' regular online SPIN Cohort assessments. Enrollment in the feasibility trial started on June 1, 2017 and was completed on June 18, 2017 when 40 eligible SPIN Cohort participants were randomized. Of these, 24 (60%) were allocated to the SPIN-HAND arm, and 16 (40%) to the usual care arm.
Period: Overall Study
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Started | 24 | 16
Completed | 24 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.5) | 58.7 (16.8) | 57.8 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 12 | 34
  Black | 1 | 2 | 3
  Other | 1 | 2 | 3
Education [Mean (Standard Deviation); unit: years] | 15.0 (3.2) | 15.2 (3.1) | 15.1 (3.1)
Married or living as married [Count of Participants; unit: Participants] | 17 | 10 | 27
Country [Count of Participants; unit: Participants]
  Canada | 8 | 4 | 12
  United States | 9 | 7 | 16
  United Kingdom | 7 | 5 | 12
Time since onset first non-Raynaud's symptom or sign [Mean (Standard Deviation); unit: years] — Population: Please note that there is some missing data on some disease characteristics for some participants
  years
    number analyzed (Participants) | 24 | 14 | 38
    (all) | 11.8 (7.0) | 11.6 (9.5) | 11.7 (7.9)
Time since onset Raynaud's [Mean (Standard Deviation); unit: years] — Population: Please note that there is data missing on some of the disease characteristics for some participants.
  years
    number analyzed (Participants) | 23 | 14 | 37
    (all) | 14.6 (11.2) | 15.7 (13.6) | 15.0 (12.0)
Time since diagnosis [Mean (Standard Deviation); unit: years] — Population: Please note that there is data missing on some of the disease characteristics for some participants.
  years
    number analyzed (Participants) | 24 | 15 | 39
    (all) | 10.0 (6.2) | 10.1 (8.3) | 10.1 (7.0)
Diffuse disease subtype [Count of Participants; unit: Participants] | 11 | 8 | 19
Modified Rodnan Skin Score [Mean (Standard Deviation); unit: scores on a scale] — The Modified Rodnan Skin Score (mRSS) is used to measure skin thickness in clinical trials of systemic sclerosis. An examiner pinches the skin slightly in 17 different areas on the patient and gives a score ranging from 0-3 assessing the patients skin thickness as; normal, no skin thickness (mRSS= 0), mild (mRSS =1), moderate (mRSS= 2), and severe (mRSS=3). These scores (0-3) are applied to each of the 17 areas, therefore total scores range from 0 to 51. Population: Please note that there is data missing on some of the disease characteristics for some participants.
  scores on a scale
    number analyzed (Participants) | 20 | 11 | 31
    (all) | 9.7 (10.8) | 17.4 (10.8) | 12.4 (11.2)
Small joints contractures [Count of Participants; unit: Participants] — Proportion of participants with small joint contractures (% positive)
  Participants | 6 | 7 | 13
Large joint contractures [Count of Participants; unit: Participants] — Proportion of participants with large joint contractures (% positive)
  Participants | 4 | 4 | 8
Tendon friction rubs [Count of Participants; unit: Participants] — Proportion of participants with tendon friction rubs (% positive) Population: Please note that there is data missing on some of the disease characteristics for some participants.
  Participants
    number analyzed (Participants) | 23 | 11 | 34
    (all) | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Eligibility: Number of Patients in the SPIN Cohort Who Meet the Cut-off Thresholds for Eligibility
Description: Measure: count of eligible patients
Time Frame: baseline
Population: Enrollment in the feasibility trial started on June 1, 2017 and was completed on June 18, 2017 when 40 eligible SPIN Cohort participants were randomized. Of these, 24 (60%) were allocated to the SPIN-HAND arm, and 16 (40%) to the usual care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
Participants | 24 | 16

2. Primary Outcome: Enrolment: Percentage of Patients Who Consent to Participation
Description: Measure: count of consenting patients
  Participants randomized to be offered the intervention received an automated email invitation including a link to the SPIN-HAND Program site and the consent form for the intervention. Participants who were randomized to care as usual were not notified that they had not been offered the intervention and completed their regular SPIN Cohort assessments. Thus, participants who were offered the intervention were not blind to their status, whereas participants assigned to usual care were blind to their participation in the trial and to their assignment to usual care.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
Participants | 15 | 0

3. Primary Outcome: Participant Grade on Usability of the SPIN-HAND Program Based on Post-trial Patient Interviews
Description: At 3-months post-randomization, qualitative semi-structured interviews were conducted with participants in the intervention arm to assess user acceptability and satisfaction. The interview, consisting of 29 questions, was guided by items of the Patient Education Materials Assessment Tool for Audiovisual Materials and addressed topics related to usability, understandability, organization, and clarity. During these interviews, participants were asked to give the SPIN-HAND program a grade ranging from 0-10, 0 being the worst and 10 being the best possible score. In this table, we report the overall mean grade reported by the intervention arm participants who agreed to be interviewed post-trial.
Time Frame: 3 months
Population: Of the 15 intervention arm participants, 6 participated in the interview. Of the 9 participants who were not interviewed, 1 withdrew a few days after consenting to the feasibility trial, 3 were unreachable at 3-month post-randomization (3 contact attempts), 5 declined (2 participants indicated that they did not use the program enough, 2 declined due to health problems, 1 mentioned exercise was not a priority). None of the participants randomized to usual care participated in these interviews.
Measure: Mean (Standard Deviation); unit: Overall mean grade for SPIN-HAND program
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 6 | 0
Overall mean grade for SPIN-HAND program | 8.5 (1.5) |

4. Primary Outcome: Intervention Use: Number of Logins to the SPIN-HAND Program and Number of Participants Who Accessed SPIN-HAND Program Online Features
Description: Usage of the online SPIN-HAND program was measured based on usage log data, notably the number of participants who logged into the program once, twice or more than two times. Program usage was also measured based on the number of participants who accessed different parts of the online SPIN-HAND program including: the introduction videos, the website tour, the page explaining the level of hand involvement to identify the exercises most relevant to them, the four available modules of the online SPIN-HAND program, as well as the goal-setting feature.
Time Frame: 3 months
Population: None of the participants randomized to usual care logged into the SPIN-HAND program.
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 15 | 0
Participants
  Logged in 1 time | 7 |
  Logged in 2 times | 3 |
  Logged in more than 2 times | 5 |
  Number of participants who watched introduction videos | 11 |
  Number of participants who used the website tour | 6 |
  Number of participants who accessed page to identify relevant exercises | 10 |
  Number of participants who did not access any module | 6 |
  Number of participants who accessed 1 of the 4 modules | 4 |
  Number of participants who accessed 3-4 modules | 2 |
  Number of participants who used the goal-setting feature | 4 |

5. Primary Outcome: Usage Log Data: Completeness of the Automatic Usage Log Data Values Collected
Description: Here we report our success in collecting participant usage log data. This is reported as the percentage of the usage log data that was successfully collected.
Time Frame: 3 months
Population: None of the participants randomized to usual care logged into the SPIN-HAND program
Measure: Number; unit: Percent completeness of usage log data
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 15 | 0
Percent completeness of usage log data | 100 |

6. Primary Outcome: Usage Log Data: Linking of Data From the SPIN Cohort and SPIN-HAND Platforms.
Description: We report our percentage success in linking data coming from the SPIN Cohort and SPIN-HAND platforms.
Time Frame: 3 months
Population: None of the participants randomized to usual care logged into the SPIN-HAND program
Measure: Number; unit: % success linking participant data
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 15 | 0
% success linking participant data | 100 |

7. Primary Outcome: Count of Participants Who Reported Technological Problems During Post-trial Patient Interviews
Description: Measure: count of technological problems reported
  SPIN personnel reported no issues with the technological performance of the online SPIN-HAND program. As part of the user feedback interviews, participants of the SPIN-HAND program were asked whether they experienced technological difficulties during the intervention. Here, we report the number of intervention-arm participants who reported technological issues, during these post-trial interviews. In cases of technological difficulty experienced by participants, technological assistance was provided by the SPIN team, and the issues were resolved.
Time Frame: 3 months
Population: 6 of the 15 intervention arm participants agreed to be interviewed post-trial. Participants randomized to usual care were not interviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 6 | 0
Participants
  Participants who reported no technology issues | 4 | 0
  Participants who reported internet connectivity issues | 1 |
  Participants who reported login issue (resolved by SPIN team) | 1 |

8. Secondary Outcome: The Cochin Hand Function Scale (CHFS)
Description: The Cochin Hand Function Scale (CHFS) measures functional ability of the hand among patients with rheumatic diseases. The 18-item CHFS measures ability to perform daily hand-related activities (e.g., kitchen, dressing oneself, hygiene, writing/typing). Items are scored on a 0-5 Likert scale (0=without difficulty; 5=impossible). Higher scores indicate less functionality. The total score is obtained by adding the scores of all items (range 0-90).
Time Frame: Baseline, 3 months
Population: Of the 40 participants, 26 (65%) completed their 3-months follow-up assessments, including 14 in the intervention arm (58%) and 12 in the control arm (75%).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
units on a scale
  Baseline | 21.9 (15.5) | 21.1 (16.1)
  Month 3: number analyzed (Participants) | 14 | 12
  Month 3 | 22.0 (15.5) | 20.9 (6.6)

9. Secondary Outcome: EuroQol Group 5 Dimension 5 Level (EQ-5D-5L): Number of Participants Per Dimension Per Level
Description: The EuroQol Group 5 Dimension 5 Level (EQ-5D-5L) is standardized questionnaire measuring 5 dimensions related to health related quality of life, mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, items are rated from 1 (no problems) to 5 (extreme problems). Here we report the number of intervention arm and control arm participants who gave scores ranging 1-5 for the different dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), at baseline and at 3-months post randomization.
Time Frame: Baseline, 3 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
Participants
  Mobility - Baseline: Level 1 | 7 | 5
  Mobility - Baseline: Level 2 | 8 | 6
  Mobility - Baseline: Level 3 | 8 | 3
  Mobility - Baseline: Level 4 | 1 | 2
  Mobility - Baseline: Level 5 | 0 | 0
  Mobility - Month 3: number analyzed (Participants) | 14 | 12
  Mobility - Month 3: Level 1 | 5 | 7
  Mobility - Month 3: Level 2 | 7 | 1
  Mobility - Month 3: Level 3 | 0 | 2
  Mobility - Month 3: Level 4 | 2 | 2
  Mobility - Month 3: Level 5 | 0 | 0
  Self care - Baseline: Level 1 | 10 | 7
  Self care - Baseline: Level 2 | 9 | 7
  Self care - Baseline: Level 3 | 4 | 1
  Self care - Baseline: Level 4 | 0 | 1
  Self care - Baseline: Level 5 | 1 | 0
  Self care - Month 3: number analyzed (Participants) | 14 | 12
  Self care - Month 3: Level 1 | 8 | 4
  Self care - Month 3: Level 2 | 3 | 7
  Self care - Month 3: Level 3 | 2 | 1
  Self care - Month 3: Level 4 | 1 | 0
  Self care - Month 3: Level 5 | 0 | 0
  Usual activity - Baseline: Level 1 | 6 | 0
  Usual activity - Baseline: Level 2 | 8 | 8
  Usual activity - Baseline: Level 3 | 8 | 5
  Usual activity - Baseline: Level 4 | 2 | 3
  Usual activity - Baseline: Level 5 | 0 | 0
  Usual activity - Month 3: number analyzed (Participants) | 14 | 12
  Usual activity - Month 3: Level 1 | 4 | 2
  Usual activity - Month 3: Level 2 | 6 | 5
  Usual activity - Month 3: Level 3 | 2 | 4
  Usual activity - Month 3: Level 4 | 2 | 1
  Usual activity - Month 3: Level 5 | 0 | 0
  Pain/Discomfort - Baseline: Level 1 | 2 | 1
  Pain/Discomfort - Baseline: Level 2 | 10 | 4
  Pain/Discomfort - Baseline: Level 3 | 9 | 8
  Pain/Discomfort - Baseline: Level 4 | 3 | 3
  Pain/Discomfort - Baseline: Level 5 | 0 | 0
  Pain/Discomfort - Month 3: number analyzed (Participants) | 14 | 12
  Pain/Discomfort - Month 3: Level 1 | 1 | 0
  Pain/Discomfort - Month 3: Level 2 | 5 | 2
  Pain/Discomfort - Month 3: Level 3 | 5 | 10
  Pain/Discomfort - Month 3: Level 4 | 3 | 0
  Pain/Discomfort - Month 3: Level 5 | 0 | 0
  Anxiety/Depression - Baseline: Level 1 | 8 | 5
  Anxiety/Depression - Baseline: Level 2 | 11 | 8
  Anxiety/Depression - Baseline: Level 3 | 3 | 3
  Anxiety/Depression - Baseline: Level 4 | 2 | 0
  Anxiety/Depression - Baseline: Level 5 | 0 | 0
  Anxiety/Depression - Month 3: number analyzed (Participants) | 14 | 12
  Anxiety/Depression - Month 3: Level 1 | 11 | 6
  Anxiety/Depression - Month 3: Level 2 | 2 | 4
  Anxiety/Depression - Month 3: Level 3 | 1 | 1
  Anxiety/Depression - Month 3: Level 4 | 0 | 1
  Anxiety/Depression - Month 3: Level 5 | 0 | 0

10. Secondary Outcome: EuroQol Group 5 Dimension 5 Level (EQ-5D-5L): Visual Analogue Scale (VAS) Scores for Patient Self-rated Health
Description: As part of the EQ-5D-5L questionnaire, a Visual Analogue Scale (VAS) records the patient's self-rated health on a scale from 0-100 where the endpoints are labelled 'the best health you can imagine' (100) and 'the worst health you can imagine' (0). Here we report the mean (and standard deviations) self-reported patient health VAS scores of intervention arm participants and control arm participants (i.e. usual care), at baseline and at 3-months post-randomization.
Time Frame: Baseline, 3 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
score on a scale
  Baseline | 64.9 (19.7) | 56.8 (15.9)
  Month 3: number analyzed (Participants) | 14 | 12
  Month 3 | 66.9 (19.8) | 54.9 (13.1)

11. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS-29) Profile Version 2.0
Description: Measures 8 domains of health status with 4 items for each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference) plus a single item for pain intensity. Items are scored on a 5-point scale (range 1-5), with different response options for different domains, and the single pain intensity item is measured on an 11-point rating scale. Higher scores represent more of the domain being measured; that is, better physical function and ability to participate in social roles and activities, but higher levels of anxiety, depression, fatigue, sleep disturbance, pain interference, and pain intensity. Total raw scores are obtained by summing item scores for each domain, which are converted into T-scores standardized from the general US population (mean=50, SD=10). Here, we report the pre- and post-intervention total scores for PROMIS-29 domains.
Time Frame: Baseline, 3 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
Number analyzed (Participants) | 24 | 16
T-score
  PROMIS-29 Physical Function Domain- Baseline | 40.7 (8.9) | 39.4 (6.5)
  PROMIS-29 Physical Function Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Physical Function Domain- Month 3 | 42.2 (8.6) | 41.1 (6.6)
  PROMIS-29 Anxiety Domain- Baseline | 53.8 (10.5) | 56.7 (9.9)
  PROMIS-29 Anxiety Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Anxiety Domain- Month 3 | 48.7 (8.2) | 53.2 (9.6)
  PROMIS-29 Depression Domain- Baseline | 51.8 (10.1) | 53.7 (9.9)
  PROMIS-29 Depression Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Depression Domain- Month 3 | 47.4 (8.0) | 51.6 (9.8)
  PROMIS-29 Fatigue Domain- Baseline | 58.3 (12.0) | 59.3 (7.4)
  PROMIS-29 Fatigue Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Fatigue Domain- Month 3 | 55.7 (10.7) | 58.7 (8.9)
  PROMIS-29 Sleep Domain- Baseline | 54.3 (8.7) | 53.6 (9.6)
  PROMIS-29 Sleep Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Sleep Domain- Month 3 | 50.4 (6.7) | 54.3 (6.1)
  PROMIS-29 Social Roles Domain- Baseline | 46.0 (8.7) | 42.3 (7.8)
  PROMIS-29 Social Roles Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Social Roles Domain- Month 3 | 49.5 (10.0) | 40.7 (8.2)
  PROMIS-29 Pain Interference Domain- Baseline | 57.7 (9.9) | 61.7 (5.9)
  PROMIS-29 Pain Interference Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Pain Interference Domain- Month 3 | 56.1 (7.8) | 60.6 (6.7)
  PROMIS-29 Pain Intensity Domain- Baseline | 4.7 (2.8) | 5.9 (1.9)
  PROMIS-29 Pain Intensity Domain- Month 3: number analyzed (Participants) | 14 | 12
  PROMIS-29 Pain Intensity Domain- Month 3 | 4.9 (2.7) | 5.3 (1.9)

ADVERSE EVENTS:
Time Frame: Assessed throughout the intervention period (i.e. 3-months post-randomization), and during the post-trial interviews with intervention arm participants at 3-months post-randomization
Arm/Group | SPIN-HAND Program | Not Offered the SPIN-HAND Program
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/16
Other Adverse Events (participants affected / at risk) | 0/24 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03092024/Prot_SAP_000.pdf